CLINICAL TRIAL: NCT05182528
Title: Hematological Disorders in Covid 19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa mahmoud elsayed, Dr/Radwa mahmoud elsayed, Assiut University
Other Study IDs: Hematological disorders
Record Dates: First submitted 2022-01-06; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Hematological Abnormalities in covid19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
aim of the research is to detect hematological abnormalities in covid 19 patients and its correlation with the severity and outcome of the disease.

DETAILED DESCRIPTION:
Covid 19 is an infectious disease caused by a newly discovered coronavirus.most people infected with the covid 19 virus will have mild to moderate respiratory illness and recover without specific treatment.older people and those with underlying medical problems like cardiac diseases,diabetes,any chronic respiratory disease and cancer are more likely to have serious illness.the covid 19 virus spreads primarily through droplets of saliva or discharge from the nose oral cavity when an infected person coughs or sneezes.people with covid19 have had a wide range of symptoms reported _ranging from mild to severe symptoms.symptoms may appear 2_14 days after exposure to the infection .any one can have mild to severe symptoms.people with these symptoms may have covid 19: fever or shivering,cough,shortness of breath,fatigue,body or muscle aches,headache,new loss of smell or taste ,sore thraot,congestion or running nose , nausea or vomiting,diarrhoea.

The most common hematological clinical findings include lymphocytopenia,neutrophilia,eosinophilia,mild thrombocytopenia,and less frequently thrombocytosis,the presence of reactive lymphocytes has been reported only occasionally the leucocyte count may be normal,reduced or increased.according to a meta analysis leucocytosis,lymphopenia and thrombocytopenia are associated with greater severity and fatality in covid 19 cases

ELIGIBILITY:
Inclusion Criteria:

all covid 19 patients diagnosed by pcr or CT chest

-

Exclusion Criteria:

* No

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Covid 19 patients ranging from 18 years old to 90 years old
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Hematological disorders in covid 19 patients | Baseline
  to detect hematological abnormalities in covid 19 patients and its correlation to outcome and severity of the disease

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mizurini DM, Hottz ED, Bozza PT, Monteiro RQ. Fundamentals in Covid-19-Associated Thrombosis: Molecular and Cellular Aspects. Front Cardiovasc Med. 2021 Dec 17;8:785738. doi: 10.3389/fcvm.2021.785738. eCollection 2021. PMID 34977191